CLINICAL TRIAL: NCT06724055
Title: Diagnostic Prediction of Pancreatic Masses: How to Avoid an Unnecessary Resection
Brief Title: Diagnostic Prediction of Pancreatic Masses
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-DPPM
Record Dates: First submitted 2024-11-18; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Masses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- AIP
- PPL
- PDAC

SUMMARY:
The goal of this observational study is to learn if a strategy can be developed for differentiating autoimmune pancreatitis (AIP) and primary pancreatic lymphoma (PPL) from pancreatic ductal adenocarcinoma (PDAC) in patients presenting with pancreatic masses. The main question it aims to answer is:

What features, in the perspectives of clinical manifestation, laboratory tests, and imaging, can differentiate different kinds of pancreatic masses (AIP, PPL and PDAC)?

Participants will not be given any interventions since this is a retrospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients presenting with pancreatic masses and eventually diagnosed with PPL, AIP, or PDAC (confirmed by pathologic results).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients in Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic nomogram | From date of admission into the hospital to the establishment of diagnosis, assessed up to 100 months

SECONDARY OUTCOMES:
serum level of LDH | From date of admission into the hospital to the establishment of diagnosis, assessed up to 100 months
serum level of IgG4 | From date of admission into the hospital to the establishment of diagnosis, assessed up to 100 months
largest diameter of pancreatic masses | From date of admission into the hospital to the establishment of diagnosis, assessed up to 100 months
dilation of pancreatic duct | From date of admission into the hospital to the establishment of diagnosis, assessed up to 100 months

IPD SHARING:
Plan to Share IPD: No